CLINICAL TRIAL: NCT03281811
Title: A Pilot Study of Photodynamic Therapy in Refractory Plaques and Tumors of Mycosis Fungoides
Brief Title: Photodynamic Therapy in Treating Patients With Refractory Mycosis Fungoides
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC168B; NCI-2017-01649 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC168B (Other: Mayo Clinic in Arizona)
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2021-02

CONDITIONS: Refractory Mycosis Fungoides
MeSH Terms: conditions — Mycosis Fungoides | interventions — Aminolevulinic Acid; Photochemotherapy; 1-phenyl-3,3-dimethyltriazene; Phototherapy; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (aminolevulinic acid hydrochloride, PDT, RT) (Experimental): Patients receive aminolevulinic acid hydrochloride topically and undergo photodynamic therapy on day 1. Treatment repeats every 4 weeks for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Beginning at week 24, patients undergo radiation therapy daily for 4 weeks.
  Interventions: Drug: Aminolevulinic Acid Hydrochloride; Drug: Photodynamic Therapy; Other: Quality-of-Life Assessment; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Aminolevulinic Acid Hydrochloride — Given topically
  Other Names: .delta.-Aminolevulinic acid hydrochloride; Alacare; Ameluz; Aminolevulinic Acid HCl; Delta-Aminolevulinic Acid HCl; Delta-Aminolevulinic Acid Hydrochloride; Levulan; Levulan Kerastick
Drug: Photodynamic Therapy — Undergo PDT
  Other Names: PDT; Photoradiation Therapy
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Radiation: Radiation Therapy — Undergo RT
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; irradiation; Radiation; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation

SUMMARY:
This pilot phase II trial studies how well photodynamic therapy works in treating patients with mycosis fungoides that does not respond to treatment. Photodynamic therapy uses a drug, such as aminolevulinic acid hydrochloride, that becomes active when it is exposed to light. The activated drug may kill cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy of photodynamic therapy (PDT) in refractory tumors and plaques of mycosis fungoides (MF).

SECONDARY OBJECTIVES:

I. To determine the effects of sequential PDT and radiation therapy (RT). II. To determine the side effect profile of PDT in MF.

EXPLORATORY OBJECTIVES:

I. To determine the quality of life during and after treatment.

OUTLINE:

Patients receive aminolevulinic acid hydrochloride topically and undergo photodynamic therapy on day 1. Treatment repeats every 4 weeks for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Beginning at week 24, patients undergo radiation therapy daily for 4 weeks.

After completion of study treatment, patients are followed up for up to 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of mycosis fungoides as confirmed by the Mayo Clinic Arizona Dermatopathology Department
* Patients must have a tumor or plaque that is refractory to conventional treatment including but not limited to one of the following (up to 4 lesions in a single field of PDT or RT will be considered for treatment):

  * Plaque stage disease that has failed at least 2 skin directed therapies (including topical steroids) or refractory plaques despite at least one systemic therapy or plaques with evidence of folliculotropism
  * The presence of a tumor of MF
* Negative urine pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Ability to complete questionnaire(s) by themselves or with assistance
* Provide written informed consent
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)

Exclusion Criteria:

* Prior radiation to the same site deemed to be too high of level of radiation for retreatment
* Photosensitivity disorder, including but not limited to porphyria, or concomitant photosensitizing drugs that place the patient at an elevated risk of developing severe side effects to PDT or RT
* Skin cancer other than actinic keratosis, basal cell carcinoma, and squamous cell carcinoma in situ in the field of RT
* Active infection at the site to be irradiated
* Any underlying condition which prevents the patient from being able to undergo the required number of sessions of PDT or RT and required follow up
* Pregnancy
* Lactation and a radiation field which would include the breast or nipple or deemed to place the mother or child at elevated risk of radiation exposure (evaluated by MRP, ARM, WR, WW)
* An allergy to a component of Levulan
* Women of childbearing potential (post-menopausal or not of child-bearing potential) is defined by: 1 year of natural (spontaneous) amenorrhea or surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or tubal ligation at least 6 weeks ago; oophorectomy alone must confirmed by follow up hormone level assessment to be considered not of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using basic methods of contraception which includes:

  * Total abstinence (Periodic abstinence and withdrawal are not acceptable methods of contraception)
  * Female sterilization (bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least 6 weeks before taking study treatment; oophorectomy alone requires follow up hormone level assessment for fertility
  * Male sterilization (at least 6 months prior to screening); the vasectomized male partner should be the sole partner for that subject
  * Barrier methods of contraception: condom or occlusive cap
  * Use of oral, injected or implanted hormonal methods of contraception or other forms or hormonal contraception that have complete efficacy (failure < 1%); (the dose of the contraceptive should be stable for 3 months)
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy; NOTE: Patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-08-12 (Actual)

PRIMARY OUTCOMES:
Complete clinical response | At 24 weeks
  Will be determined by Composite Assessment of Index Lesion Severity (CAILS) and Physician Global Assessment (PGA).

SECONDARY OUTCOMES:
Change in CAILS score | Baseline up to week 24
  Will be conducted and summarized using means, standard deviations and 95% confidence intervals. Statistical tests on endpoints (t-test for continuous data; Wilcoxon rank-sum test, Fisher?s exact test, or Chi-square test for ordinal data) will be utilized to determine differences at any particular time point. Graphical displays will be produced, such as mean profile plots or bar charts.
Change in field of treatment | Baseline up to week 24
  Will be conducted and summarized using means, standard deviations and 95% confidence intervals. Statistical tests on endpoints (t-test for continuous data; Wilcoxon rank-sum test, Fisher?s exact test, or Chi-square test for ordinal data) will be utilized to determine differences at any particular time point. Graphical displays will be produced, such as mean profile plots or bar charts.
Change in Skindex-16 score | Baseline up to week 24
  Will be conducted and summarized using means, standard deviations and 95% confidence intervals. Statistical tests on endpoints (t-test for continuous data; Wilcoxon rank-sum test, Fisher?s exact test, or Chi-square test for ordinal data) will be utilized to determine differences at any particular time point. Graphical displays will be produced, such as mean profile plots or bar charts.
Incidence of adverse events (AEs) | Up to 2 years
  The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. AE incidence and severity as measured by the Common Terminology Criteria for Adverse Events (CTCAE) version (v)4.0.

OTHER OUTCOMES:
Patient-reported outcomes | Up to 2 years
  Patient-reported symptoms will be described at each time point using the mean, confidence interval, median, and range. Graphical procedures will include stream plots of individual patient scores and plots of average values over time. Correlational analyses will be done to determine the relationships among patients-reported symptoms, as well as with clinical outcomes (response) and clinician-assessed symptoms (National Cancer Institute [NCI] CTCAE v4).
Quality of life (QOL) | Up to 2 years
  Patient-reported symptoms and QOL will be described at each time point using the mean, confidence interval, median, and range. Graphical procedures will include stream plots of individual patient scores and plots of average values over time. Correlational analyses will be done to determine the relationships among patients-reported symptoms and QOL, as well as with clinical outcomes (response) and clinician-assessed symptoms (NCI CTCAE v4).

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Mangold, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials